CLINICAL TRIAL: NCT00378443
Title: ACEi/ARB Alone Versus ACEi/ARB Plus Steroids in the Treatment of Primary IgA Nephropathy, a RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2006]022
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Last update posted 2006-09-22 (Estimated); Status verified 2006-09

CONDITIONS: Glomerulonephritis, IGA
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Prednisone; Cilazapril; Losartan

INTERVENTIONS:
Drug: prednisone + Inhibace/Cozaar
Drug: Inhibace/Cozaar

SUMMARY:
IgA nephropathy( IgAN) is the most common primary glomerulonephritis worldwide. Since the etiology of the disease is not clearly understood, no specific therapeutic strategies was defined for IgAN. Both ACEi/ARB and steroid was found to be effective in slowing the rate of disease progression, but the use of steroid was restricted because of its side effects. However, there is no evidence from RCT on the question of whether combined use of steroid with ACEi/ARB can bring more benefit to IgAN patients than ACEi/ARB alone. We therefore undertook a randomized, multicenter study to investigate the efficacy and safety profile of combined use of ACEi/ARB plus steroid compared with ACEi/ARB alone in the treatment of patients with IgAN.

DETAILED DESCRIPTION:
IgA nephropathy( IgAN) is the most common primary glomerulonephritis worldwide. Since the etiology of the disease is not clearly understood, no specific therapeutic strategies was defined for IgAN. In the many studies on the treatment of IgAN, both ACEi/ARB and steroid was found to be effective in slowing the rate of disease progression, but the use of steroid was restricted because of its side effects, and ACEi/ARB was considered to be the first line therapy. However, there is no evidence from RCT on the question of whether combined use of steroid with ACEi/ARB can bring more benefit to IgAN patients than ACEi/ARB alone. We therefore undertook a randomized, multicenter study to investigate the efficacy and safety profile of combined use of ACEi/ARB plus steroid compared with ACEi/ARB alone in the treatment of patients with IgAN.

ELIGIBILITY:
Inclusion Criteria:

1. underwent renal biopsy within 1 year before start fo trial;
2. 24 hour urinary protein excretion ranged between 1 to 7 g/d;
3. eGFR, evaluated by MDRD formula, should be higher than 30 ml/min

Exclusion Criteria:

1. crescentic glomerulonephritis;
2. steroid therapy subjected within 1 year before trial;
3. malignant hypertension(DBP> 130 mmHg and/or SBP> 220mmHg), resistant to anti-hypertensive agents;
4. urinary protein excretion decrease below 1 g/l after run-in period;
5. Myocardial infarction or cerebrovascular accident in 6 months preceding the trial;
6. renovascular disease;
7. diabetes mellitus;
8. Malignancy, severe liver disease, refractory infection;
9. peptic ulcer in active disease phase;
10. pregnancy;
11. other contraindication to the use of ACEi/ ARB or corticosteroid;
12. alcohol abuse or drug addiction

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-01; Study Completion 2007-06

PRIMARY OUTCOMES:
Serum creatinine
24 hour urinary protein excretion

SECONDARY OUTCOMES:
Urinalysis
serum urea
serum albumin

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, MD, Principal Investigator — Renal Division, Peking University First Hospital

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] Lv J, Zhang H, Chen Y, Li G, Jiang L, Singh AK, Wang H. Combination therapy of prednisone and ACE inhibitor versus ACE-inhibitor therapy alone in patients with IgA nephropathy: a randomized controlled trial. Am J Kidney Dis. 2009 Jan;53(1):26-32. doi: 10.1053/j.ajkd.2008.07.029. Epub 2008 Oct 19. PMID 18930568